CLINICAL TRIAL: NCT05613933
Title: Effectiveness of Antibiotic Prophylaxis of Infective Endocarditis Before Invasive Dental Procedures in Patients With Prosthetic Heart Valves and/or History of Infective Endocarditis: a Prospective, Registry-based, Cluster-randomized Trial in Primary Care
Brief Title: Effectiveness of Antibiotic Prophylaxis of Infective Endocarditis for Invasive Dental Procedures in Patients With Prosthetic Heart Valves and/or History of Infective Endocarditis
Acronym: PROPHETS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2021/24
Record Dates: First submitted 2022-02-15; First posted 2022-11-14 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Endocarditis, Bacterial; Endocarditis; Endocarditis Acute and Subacute
Keywords: Registry based randomized controlled trial; antibiotic prophylaxy; dentist; invasive dental procedure; infective endocarditis
MeSH Terms: conditions — Endocarditis, Bacterial; Endocarditis

STUDY DESIGN:
Intervention Model Description: A 2-arm, registry-based, cluster RCT, to be conducted in all French Health Territories (Territoires de santé, TDS) of metropolitan France, which will serve as randomization clusters
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): In the intervention arm, dentists will receive information on the study 8 weeks before the start of the study and will be invited to consent to participate or to opt out
  Interventions: Other: Improved practices
- Control arm (No Intervention): In the clusters randomized to the control arm, no intervention will be performed and no information will be sent to dentists.

INTERVENTIONS:
Other: Improved practices — A package of tools including: antibiotic prophylaxis guidelines reminders, periodic reminders, the Infectious Endocarditis Prevention Card for patients at risk, practical information targeting both dentists and patients, etc…
  Arms: Intervention arm

SUMMARY:
Infective endocarditis (IE) continues to cause serious morbidity and mortality. To reduce its incidence, antibiotic prophylaxis has been recommended before invasive dental procedures in patients with at risk predispositions. Several studies have examined the effect of antibiotic prophylaxis on the incidence of IE and have brought conflicting results. The investigators aim to evaluate the effectiveness of antibiotic prophylaxis before invasive dental procedures to prevent oral streptococcal infective endocarditis in patients with prosthetic heart valves and/or history of IE, using a registry-based, cluster-randomized, controlled trial. In secondary objectives, the investigators aim to analyze changes in dentists' practices.

DETAILED DESCRIPTION:
Conducting a conventional individual-based RCT to demonstrate the efficacy of antibiotic prophylaxis of IE is unfeasible and unethical but it also seems unacceptable to perpetuate potentially ineffective and ecologically deleterious antibiotic use. Since the conditions for an individual RCT are not met, the procedure performed does not directly involve the drug but rather the practices of the dentists. This trial will be based on the hypothesis that dentists of health territories (territoires de santé; TDS) allocated to the intervention arm will increase their prescription of antibiotic prophylaxis in patients with prosthetic heart valve and/or history of IE. Thus, assuming antibiotic prophylaxis is effective, the intervention arm should be associated with a decrease in the incidence of oral streptococci IE as compared to the control arm.

In the intervention arm, dentists will receive information on the study before the start of the study.Those who consent will receive information with an "antibiotic prophylaxis package" aimed to improve adherence to current guidelines. These interventions will be periodically repeated in order to ensure the persistence of their effect over time.

Among included patients, dental procedures will be classified as invasive if they imply manipulation of the gingival or periapical region of the teeth or a perforation of the oral mucosa. In these patients, exposure to antibiotic prophylaxis will be identified through the dispensation of an antibiotic treatment active against oral streptococci in the 21 days before the dental procedure. At each new invasive procedure, individuals will be followed for 3 months, until the study outcome, hospital admission for valve replacement, or death from any cause

ELIGIBILITY:
Inclusion Criteria:

* All French Health Territories (Territoires de santé, TDS) will be included and each TDS will contribute as a cluster for randomization.
* All dentists working in each TDS will be included.
* Among individuals receiving an invasive dental procedure, all patients aged 18 years or more identified with prosthetic heart valves or recorded with prior infective endocarditis will be included.

Exclusion Criteria:

* No exclusion criteria for health territories, dentists and patient.
* However, dental procedures that had been performed less than 6 months after the date of first implantation of prosthetic heart valve won't be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250000 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of infective endocarditis | Within 3 months after an invasive dental procedure
  Diagnosis of infective endocarditis due to oral streptococci that occurs within 3 months after an invasive dental procedure

SECONDARY OUTCOMES:
Antibiotic prophylaxis rate | 21 days before the dental procedure
  Antibiotic prophylaxis rate in dentists according to their randomization arm (Health territories) in all patients regardless of the implantation of prosthetic heart valve and/or history of IE and their dental procedures (invasive or not). The antibiotic prophylaxis will be classified as appropriate (following the recommendation/intervention) or inappropriate